CLINICAL TRIAL: NCT06013410
Title: Pathophysiological Effects of Persistently Colonized Microbiome on Irritable Bowel Syndrome
Acronym: IBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-0381
Record Dates: First submitted 2023-06-12; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS group (Experimental): patients diagnosed with IBS according to clinical presentations
  Interventions: Diagnostic Test: colonoscopy
- Healthy control group (No Intervention): healthy control group

INTERVENTIONS:
Diagnostic Test: colonoscopy — colonoscopy
  Arms: IBS group

SUMMARY:
The goal of this clinical trial is to explore the pathophysiological effects of the persistently colonized microbiome in irritable bowel syndrome (IBS) patients. The main questions it aims to answer are:

Question 1: the microbiome difference of the biofilm between IBS and healthy patients.

Question 2: the metabolic product patterns between IBS and healthy patients.

Participants will need to take a colonoscopy examination, two gut mucosal biopsy samples will be collected during the examination.

Researchers will compare the IBS and healthy control groups to see if there was the disease-specific pattern in the microbiome and metabolic product of the biofilm.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients with IV type; no abdominal surgery;

Exclusion Criteria:

* age <18 y;
* major disease;
* alcoholic addicted;
* antibiotic use in past 3 months;
* severe gastrointestinal disease
* severe cardiac disease;
* pregnant;
* ICU in past 1 year;
* vegeterian;
* immune disease (SLE etc.)
* mental disease;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-25 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
mirobiome difference of the fecal between IBS and health controls | Fecal samples will be collected immediately before the colonoscopy (T1) and 7 days after the colonoscopy test (T2)
  16S rDNA sequencing will be applied in fecal samples all the above participants
mirobiome difference of the fecal between IBS and health controls | Fecal samples will be collected 7 days after the colonoscopy test (T2)
  16S rDNA sequencing will be applied in fecal samples all the above participants
Metabolic changes between IBS and Healthy controls | 1 day biopsy will be collected during the colonoscopy test
  mucosal biopsy will be collected during the colonoscopy in each patients

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
share on request